CLINICAL TRIAL: NCT01789203
Title: Ciprofloxacin for Prevention of BK Infection in Renal Transplant Recipients
Brief Title: Ciprofloxacin for Prevention of BK Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Ahmed Osama Gaber, MD, Director, Houston Methodist Transplant Center, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Pro00007510; IRB0612-0114 (Other: HMRI IRB)
Record Dates: First submitted 2013-02-07; First posted 2013-02-12 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-10

CONDITIONS: BK Virus Infection
Keywords: BK infection; BK viremia; BK nephropathy; polyomavirus; fluoroquinolone; ciprofloxacin
MeSH Terms: interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ciprofloxacin (Active Comparator): Ciprofloxacin will be administered as two-250 mg capsules, administered once daily for 3 months post-transplant
  Interventions: Drug: Ciprofloxacin
- Placebo (Placebo Comparator): Matching placebo will be administered as two-capsules given once daily for 3 months post-transplant
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ciprofloxacin — Patients will be randomized 2:1 active comparator, Cipro, to placebo comparator.
  Other Names: Cipro
  Arms: Ciprofloxacin
Drug: placebo — Patients will be randomized 2:1 placebo comparator to active comparator, Cipro.
  Other Names: inactive drug; innocuous medication
  Arms: Placebo

SUMMARY:
BK infection is an important cause of graft dysfunction and graft loss after renal transplantation. It has been widely accepted that emergence of BK virus correlates with the more potent immunosuppressive agents used to lower acute rejection rates. In contrast to other opportunistic infections after transplantation, for which routine prophylactic agents are administered, there is no effective agent for the prevention of BK infection. Some data, however, suggests that quinolone antibiotics such as ciprofloxacin may have activity against BK virus. This has led us to investigate whether routine, short-term ciprofloxacin administration post-transplant can lower the incidence of BK infection.

DETAILED DESCRIPTION:
BK virus is a member of the virus family polyomaviridae ("polyoma"). The virus, which can manifest as a viral nephritis, was first described in a renal transplant recipient in 1971, however it was not until the past decade that infection with BK virus became known as an important contributor to graft dysfunction and graft loss after renal transplantation. It has been widely accepted that emergence of BK virus correlates with the more potent immunosuppressive agents currently used to lower acute rejection rates. In contrast to other opportunistic infections after transplantation, for which routine prophylactic agents are administered, there is no effective agent for the prevention of BK infection, nor is there an effective agent for treating BK infection once it occurs.

Ciprofloxacin is a well known anti-infective agent in the fluoroquinolone class of antibiotics. It is most active against gram-negative enteric pathogens, and is commonly used for a variety of infectious indications.

Though classified as antibacterial agents, fluoroquinolones have been suggested to exhibit anti-BK viral effects by interfering with helicase activity of the BK virus large T antigen. Ciprofloxacin has been shown in previous studies to reduce urine BK viral load, and BK-associated hemorrhagic cystitis in the stem cell transplant population. Ciprofloxacin has also been associated with a lower incidence of BK viremia in one retrospective study in kidney transplant recipients. Based on these reports, the investigators hope to find a reduction BK viremia and BK nephropathy using a prospective, randomized study design.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects over the age of 18 years
* Recipients of a primary or repeat renal allograft either alone (from a deceased or living donor) or as a dual-kidney transplant
* Signed informed consent form prior to any research assessment

Exclusion Criteria:

* Patients with known severe allergy to ciprofloxacin
* History of tendon rupture or tendinitis
* Use of antiarrythmic drugs known to prolong the QT interval such as class IA antiarrhythmic drugs (e.g. quinidine, procainamide, disopyramide), class III antiarrhythmic drugs (e.g. amiodarone, sotalol)
* Patients with history of previous non-renal transplantation
* Recipients administered rituximab within one year prior to transplantation, or recipients expected to receive rituximab as part of desensitization strategy or for the presence of historical donor specific antibodies
* QTc interval interval of greater than 500 msec on admission or post-operative EKG
* BK nephropathy with previous transplant
* BK viremia on admission
* Any condition present during the initial transplant hospitalization that in the investigator's judgment would increase the risk associated with participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samir J Patel, Pharm.D., Study Chair — Clinical Pharmacist; Ahmed O Gaber, MD, Principal Investigator — Director, Houston Methodist Transplant Center
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Brennan DC, Agha I, Bohl DL, Schnitzler MA, Hardinger KL, Lockwood M, Torrence S, Schuessler R, Roby T, Gaudreault-Keener M, Storch GA. Incidence of BK with tacrolimus versus cyclosporine and impact of preemptive immunosuppression reduction. Am J Transplant. 2005 Mar;5(3):582-94. doi: 10.1111/j.1600-6143.2005.00742.x. PMID 15707414
- [Background] Ali SH, Chandraker A, DeCaprio JA. Inhibition of Simian virus 40 large T antigen helicase activity by fluoroquinolones. Antivir Ther. 2007;12(1):1-6. PMID 17503741
- [Background] Leung AY, Chan MT, Yuen KY, Cheng VC, Chan KH, Wong CL, Liang R, Lie AK, Kwong YL. Ciprofloxacin decreased polyoma BK virus load in patients who underwent allogeneic hematopoietic stem cell transplantation. Clin Infect Dis. 2005 Feb 15;40(4):528-37. doi: 10.1086/427291. Epub 2005 Jan 21. PMID 15712075
- [Background] Miller AN, Glode A, Hogan KR, Schaub C, Kramer C, Stuart RK, Costa LJ. Efficacy and safety of ciprofloxacin for prophylaxis of polyomavirus BK virus-associated hemorrhagic cystitis in allogeneic hematopoietic stem cell transplantation recipients. Biol Blood Marrow Transplant. 2011 Aug;17(8):1176-81. doi: 10.1016/j.bbmt.2010.12.700. Epub 2010 Dec 23. PMID 21185389
- [Background] Gabardi S, Waikar SS, Martin S, Roberts K, Chen J, Borgi L, Sheashaa H, Dyer C, Malek SK, Tullius SG, Vadivel N, Grafals M, Abdi R, Najafian N, Milford E, Chandraker A. Evaluation of fluoroquinolones for the prevention of BK viremia after renal transplantation. Clin J Am Soc Nephrol. 2010 Jul;5(7):1298-304. doi: 10.2215/CJN.08261109. Epub 2010 May 27. PMID 20507960
- [Derived] Wajih Z, Karpe KM, Walters GD. Interventions for BK virus infection in kidney transplant recipients. Cochrane Database Syst Rev. 2024 Oct 9;10(10):CD013344. doi: 10.1002/14651858.CD013344.pub2. PMID 39382091
- [Derived] Patel SJ, Knight RJ, Kuten SA, Graviss EA, Nguyen DT, Moore LW, Musick WL, Gaber AO. Ciprofloxacin for BK viremia prophylaxis in kidney transplant recipients: Results of a prospective, double-blind, randomized, placebo-controlled trial. Am J Transplant. 2019 Jun;19(6):1831-1837. doi: 10.1111/ajt.15328. Epub 2019 Apr 4. PMID 30811872

RESULTS

PARTICIPANT FLOW:
Groups:
- Ciprofloxacin: Ciprofloxacin will be administered as two-250 mg capsules, administered once daily for 3 months post-transplant
  Ciprofloxacin: Patients will be randomized 2:1 active comparator to placebo comparator.
- Placebo: Matching placebo will be administered as two-capsules given once daily for 3 months post-transplant
  placebo
Period: Overall Study
Arm/Group | Ciprofloxacin | Placebo
Started | 133 | 67
Completed | 124 | 63
Not Completed | 9 | 4
Not completed — Adverse Event | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Death | 1 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Other | 1 | 1
Not completed — patient non-adherent | 2 | 0

BASELINE CHARACTERISTICS:
Population: Analysis performed on IIT patients (all randomized patients)
Groups:
- Total: Total of all reporting groups
Arm/Group | Ciprofloxacin | Placebo | Total
Number analyzed (Participants) | 133 | 67 | 200
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [40 to 58] | 44 [37 to 57] | 48 [39 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 20 | 74
  Male | 79 | 47 | 126
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 10 | 7 | 17
  Black or African American | 32 | 14 | 46
  Hispanic or Latino | 34 | 17 | 51
  White | 57 | 28 | 85
  Other or Unknown | 0 | 1 | 1
Repeat Transplant [Count of Participants; unit: Participants] | 10 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Developing BK Infection at 6 Months Post-transplant
Description: Number of patients (followed by proportion) developing BK infection at 6 months post-transplant. BK infection is defined as the presence of a detectable BK viral load in plasma by polymerase chain reaction (PCR), or the presence of BK viral inclusions on kidney biopsy specimens.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 133 | 67
Participants | 25 | 5

2. Secondary Outcome: Number of Patients With Gram Negative Urinary Tract Infections at 6 Months
Description: Number of patients with gram negative urinary tract infections as defined by a midstream urine sample containing 10^4 or more colony-forming units per mL
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 133 | 67
Participants | 17 | 14

3. Secondary Outcome: Number of Patients With Bacteremia at 6 Months
Description: Number of patients with bacteremic infection at 6 months. Bacteremia defined by a single positive blood culture that was not thought to be contaminated.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 133 | 67
Participants | 3 | 2

4. Secondary Outcome: Number of Patients With Quinolone-resistant Infection at 6 Months
Description: Number of patients with quinolone-resistant gram negative bacterial infections, among those with a gram-negative infection
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 18 | 14
Participants | 15 | 7

5. Secondary Outcome: Clostridium Difficile at 6 Months
Description: Clostridium difficile infection at 6 months
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 133 | 67
Participants | 1 | 0

6. Secondary Outcome: Serious Adverse Events
Description: Serious adverse events collected for up to 4 months (3 months on study drug plus 1 additional month)
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 133 | 67
Participants | 35 | 18

7. Secondary Outcome: Time to BK Infection
Description: Median time to initial BK viremia episode, days
Time Frame: 12 months
Population: Included 31 ciprofloxacin and 8 placebo patients who became BK viremic during the first 12 months
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 31 | 8
days | 90 [59 to 160] | 76.5 [59 to 295]

8. Secondary Outcome: BK Viremia at 1 Year
Description: Proportion of patients developing BK viremia at 1 year
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 133 | 67
Participants | 31 | 8

9. Secondary Outcome: First Plasma Viral Loads
Description: First BK plasma viral loads
Time Frame: 12 months
Population: included 31 ciprofloxacin and 8 placebo patients who became BK viremic during the first year
Measure: Median (Inter-Quartile Range); unit: copies/mL
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 31 | 8
copies/mL | 2514 [796 to 8754] | 1423 [724 to 19619]

10. Secondary Outcome: Acute Rejection at 1 Year
Description: Number of patients with biopsy-proven acute rejection of the allograft at 1 year, based on Banff classification
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 133 | 67
Participants | 14 | 7

11. Other Pre Specified Outcome: Graft Loss at 1 Year
Description: kidney failure within first 1 year of transplant
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 133 | 67
Participants | 14 | 7

12. Other Pre Specified Outcome: Death at 1 Year
Description: Patient death at 1 year
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ciprofloxacin | Placebo
Number analyzed (Participants) | 133 | 67
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events were collected out through 4 months (3 months of study drug administration + 1 month post- administration). Patients were asked during clinic visits to report any potential ciprofloxacin adverse event from a list of common adverse effects. Additional AEs were collected if reported by clinician. Graft loss and patient death were additionally collected out through 1 year
Arm/Group | Ciprofloxacin | Placebo
All-Cause Mortality (participants affected / at risk) | 1/133 | 1/67
Serious Adverse Events (participants affected / at risk) | 35/133 | 18/67
Other Adverse Events (participants affected / at risk) | 108/133 | 55/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ciprofloxacin (N=133) | Placebo (N=67)
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Acute kidney injury (Renal and urinary disorders) | 8 | 4
Anemia (Blood and lymphatic system disorders) | 0 | 1
Ascites (General disorders) | 0 | 1
Clostridium difficile (Infections and infestations) | 1 | 0
Chest pain (General disorders) | 1 | 0
Cytomegalovirus (Infections and infestations) | 0 | 1
Dehydration (General disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 3 | 4
Dyspnea (General disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 1 | 0
Epistaxis (General disorders) | 1 | 0
Fever (General disorders) | 1 | 2
GI bleed (Gastrointestinal disorders) | 1 | 0
Hematoma (Surgical and medical procedures) | 1 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Hyperglycemia (Endocrine disorders) | 2 | 2
Hyperkalemia (General disorders) | 1 | 0
Hypertension (Cardiac disorders) | 0 | 1
Infection (Infections and infestations) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
malignant hypertension (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pain (Gastrointestinal disorders) | 1 | 0
Nonfunctinal nephrostomy tube (Renal and urinary disorders) | 1 | 0
Radial nerve palsy (Nervous system disorders) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Small bowel obstruction (Gastrointestinal disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Urinary leak (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 4
Viral syndrome (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
VTE (Vascular disorders) | 5 | 0
Wound infection/complication (Surgical and medical procedures) | 3 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ciprofloxacin (N=133) | Placebo (N=67)
Constipation (Gastrointestinal disorders) | 12 | 3
Diarrhea (Gastrointestinal disorders) | 11 | 7
Dyspepsia (Gastrointestinal disorders) | 11 | 6
Edema (General disorders) | 15 | 13
Headache (General disorders) | 7 | 1
Hematuria (Renal and urinary disorders) | 2 | 4
Hypomagnesemia (General disorders) | 8 | 0
Insomnia (General disorders) | 8 | 3
Nausea (Gastrointestinal disorders) | 7 | 5
Osteopenia/osteoperosis (Musculoskeletal and connective tissue disorders) | 19 | 7
Proteinuria (Renal and urinary disorders) | 12 | 4
Urinary tract infections (Infections and infestations) | 18 | 15
Weight gain (General disorders) | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/03/NCT01789203/Prot_SAP_000.pdf